CLINICAL TRIAL: NCT05269576
Title: Clinical Simulation as a Learning Tool in Medical Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Fernando Martinez-Lopez, MD. Principal investigator. Anesthesiology coordinator., Corporacion Parc Tauli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FMartinez medical simulation
Record Dates: First submitted 2022-02-13; First posted 2022-03-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Simulation; Students, Medical; Feedback; Competency-based Education; Learning

STUDY DESIGN:
Masking Description: The investigator and the outcomes assessor didn't know the moment of the interventions in each participant of the group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm that receive two different interventions (clinical practice and clinical simulation). (Experimental): An analysis is carried out to the entire group prior to intervention. A second analysis is carried out to the entire group after one of the two interventions. Finally, a last analysis is carried out to the entire group after complete both types of interventions.
  We apply the study in a group of medicine students of 3rth course of the degree. We examine their competencies at the beginning of the course. Re-examination is done after they do a period of clinical practice or a period of clinical simulation. At the end of the course, all the students done both interventions (clinical practice and clinical simulation), moment when we do the last examination of their competencies.
  Interventions: Other: Clinical practice; Other: Clinical simulation

INTERVENTIONS:
Other: Clinical practice — Period of 5 days where medical students carry out hospital clinical practices with real patients supervised by professionals who teach them at the same time.
Other: Clinical simulation — Clinical simulation classes through 2 sessions of 5 simulated cases each day. All students actively participate in one or two of the simulation cases and observed and discussed all the cases in the debriefings of all of them.

SUMMARY:
The hypothesis of our work is that with the simulation techniques applied in the Medical School of the Autonomous University of Barcelona (UAB), students accelerate the learning curve of clinical skills, acquire transversal skills in medicine, and obtain a higher quality learning.

DETAILED DESCRIPTION:
Learning through simulation lies in the recreation of a clinical event, skills or techniques in the most reliable way in order to ensure a much more active experiential learning method than the traditional one built through theoretical classes.

Simulation provides the possibility of scheduling the acquisition of knowledge and skills in a safe environment, in which mistakes have no consequences, at a time and place.

The true learning of the student is significant when there is a reflection and assimilation of what he has learned.

At the Medicine School of Autonomous University of Barcelona (UAB), simulation has begun to be applied as a learning method at different times during the academic year.

The hypothesis of our work is that with the simulation techniques applied in the Medical School of the UAB, students accelerate the learning curve of clinical skills, acquire transversal skills in medicine, and obtain a higher quality learning.

The investigators have designed a prospective and descriptive study, which includes simulation analysis in 3rd year medicine students at the UAB during the academic years 2020/2021 and 2021/2022.

The main objective is to know the effectiveness of simulation in 3rd year medical students, through the objective evaluation of clinical and transversal competences with Mini Clinical Evaluation Exercise (Mini-CEX)

The secondary objectives are:

* To know the effect of clinical care practice in 3rd year medical students
* To compare the effect of simulation with that of clinical practice
* Qualitative analysis of the simulation by analyzing its objectives
* Contrast the evaluation of the objectives between student who did the simulation, observer students and teacher.
* Contrast the evaluation of the objectives between the different cases of each session
* Analysis of emotional interference in the evaluation of objectives
* To evaluate the quality of the clinical simulation

The study consists of analyzing the basic skills of medical students through a Mini Clinical Evaluation Exercise (Mini-CEX), which is carried out in three moments of the academic year:

* At the beginning, where the students have not had any previous experience with clinical practices or simulation.
* In the middle of the course, where there are two groups of students, one that has only done clinical practice and the other that has only done simulation. So an evaluation with Mini-CEX is carried out having performed only one of the two interventions.
* At the end of the course, where all the students have carried out clinical practices and simulation.

In each simulation session, 5 clinical cases are carried out, where the acquisition of the objectives of the simulation session and the emotional state of the student who is performing the simulation in the practical scenario are evaluated.

This evaluation is carried out by means of a questionnaire that is filled out for each of the cases, specifying who fills it out: the student who has carried out the simulation, the observer students or the teacher.

At the end of the simulation period, a satisfaction questionnaire is collected and answered by all the participants to assess the quality of the simulation classes.

Statistical analysis:

Mini-CEX can be evaluated using a scale from 0 to 10 in different domains. The domains are: history, physical examination, professionalism, clinical judgment, communication skills, and organization and efficiency. There is a summary domain that is the examiner's global assessment. This scale can be easily measured using a visual analog scale (VAS), as well as a 10-point Likert scale. To facilitate the power and ease of statistical calculations, the investigators will use the VAS scale as the measurement element.

There is also a categorical option in the Mini-CEX evaluation where the exam can be unsatisfactory, satisfactory or superior.

The objectives of the simulation can be evaluated using a VAS scale from 0 to 10 in different domains and a categorical option between objective achieved, partially achieved and not achieved. The domains are: history, physical examination, doctor-patient relationship and clinical judgment.

The satisfaction questionnaire can be evaluated using a scale from 0 to 5 in different questions.

Quantitative variables will be described as meas and 95% confidence interval. Qualitative variables will be described as percentages and 95% confidence interval.

Comparisons between different means will be made using t student. Comparisons between different percentages will be made using chi squared. Comparisons between different categorical variables will be made using Mantel-Haenszel test. In all cases, the investigators will use an alfa value of 0.05.

To calculate the number of students needed to calculate two means (VAS values between 0 and 10), the investigators assume a standard deviation in both means of 2 with a minimum magnitude of the effect to be detected equal to 1, an alpha error of 0.05 and a beta error of 0.05. from 0.2; the number needed for a bilateral contrast test is 63.

ELIGIBILITY:
Inclusion Criteria:

- Students in the 3rd year of medicine at the UAB (Autonomous University of Barcelona) who, at the beginning of the study, have not carried out any type of hospital clinical practice or clinical simulation.

Exclusion Criteria:

* Students with prior experience in hospital clinical practice or clinical simulation
* Students who have not attended clinical practices or simulation classes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-09-12 (Actual); Primary Completion 2022-06-22 (Estimated); Study Completion 2022-09-22 (Estimated)

PRIMARY OUTCOMES:
to know the effectiveness of simulation in 3rd year medical students, through the objective evaluation of clinical and transversal competences with Mini Clinical Evaluation Exercise (Mini-CEX) | Through study completion, an average of 6 months.
  Evaluation of competencies through Mini-CEX, which is done in 3 different moments of each course: at the beginning; after clinicar care practice or simulation session; and at the end of the course after clinical care practice and simulation session.

SECONDARY OUTCOMES:
To know the effect of clinical care practice in 3rd year medical students | Through study completion, an average of 6 months.
  Evaluation of competencies through Mini-CEX, which is done in 3 different moments of each course: at the beginning; after clinicar care practice or simulation session; and at the end of the course after clinical care practice and simulation session.
To compare the effect of simulation with that of clinical practice | Through study completion, an average of 6 months.
  Evaluation of competencies through Mini-CEX, which is done in 3 different moments of each course: at the beginning; after clinicar care practice or simulation session; and at the end of the course after clinical care practice and simulation session.
Qualitative analysis of the simulation by analyzing its objectives by questionnaire | Through study completion, an average of 6 months.
  Questionnaire to assess the achievement of the objectives of the simulation sessions (medical history, physical examination, doctor-patient relationship and correct diagnosis) and the emotional state of the participant in the scenario of simulation (nervousness and comfort). In each simulation session, we evaluated each case with this questionnaire that had to be answered by the student who did the simulation, the observer students and the teacher. The questionnaire had a categorical evaluation (achieved, partially achieved or non achieved) for every teaching objective.
Contrast the evaluation of the objectives between student who did the simulation, observer students and teacher, by questionnaire | Through study completion, an average of 6 months.
  Questionnaire to assess the achievement of the objectives of the simulation sessions (medical history, physical examination, doctor-patient relationship and correct diagnosis) and the emotional state of the participant in the scenario of simulation (nervousness and comfort). In each simulation session, we evaluated each case with this questionnaire that had to be answered by the student who did the simulation, the observer students and the teacher. The questionnaire had a categorical evaluation (achieved, partially achieved or non achieved) for every teaching objective.
Contrast the evaluation of the objectives between the different cases of each session by questionnare | Through study completion, an average of 6 months.
  Questionnaire to assess the achievement of the objectives of the simulation sessions (medical history, physical examination, doctor-patient relationship and correct diagnosis) and the emotional state of the participant in the scenario of simulation (nervousness and comfort). In each simulation session, we evaluated each case with this questionnaire that had to be answered by the student who did the simulation, the observer students and the teacher. The questionnaire had a categorical evaluation (achieved, partially achieved or non achieved) for every teaching objective; and a numerical evaluation with a visual analog scale from 0 to 10 for every teaching objective and the emotional state.
Analysis of emotional interference in the evaluation of objectives by visual analog scale | Through study completion, an average of 6 months.
  The emotional state of the participant in the scenario of simulation (nervousness and comfort) was evaluated in each case with a numerical evaluation by a visual analog scale from 0 to 10. VSA had to be answered by the student who did the simulation, the observer students and the teacher.
To evaluate the quality of the clinical simulation | Through study completion, an average of 6 months.
  Quality and satisfaction survey of the clinical simulation carried out by the participants at the end of the simulation. The investigators used a validated survey with 11 questions evaluated numerically from 1 to 5 (1 very disagree and 5 very agree).
Numerical analysis of the simulation by analyzing its objectives by visual analog scale | Through study completion, an average of 6 months.
  Numerical evaluation with a visual analog scale from 0 to 10 for every teaching objective.
Contrast the evaluation of the objectives between student who did the simulation, observer students and teacher, by visual analog scale | Through study completion, an average of 6 months.
  Numerical evaluation with a visual analog scale from 0 to 10 for every teaching objective by the student who did the simulation, the observer students and the teacher.
Contrast the evaluation of the objectives between the different cases of each session by visual analog scale | Through study completion, an average of 6 months.
  Numerical evaluation with a visual analog scale from 0 to 10 for every teaching objective in each case of the session of simulation.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Martínez-López, MD, Principal Investigator — Universitat Autonoma de Barcelona
Locations (1):
- Autonomous University of Barcelona, Bellaterra, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
At the moment, there is no project to share the study data. We are open to doing it so as soon as we see possibilities of working together with other similar groups.

REFERENCES:
- [Result] McGaghie WC, Issenberg SB, Cohen ER, Barsuk JH, Wayne DB. Does simulation-based medical education with deliberate practice yield better results than traditional clinical education? A meta-analytic comparative review of the evidence. Acad Med. 2011 Jun;86(6):706-11. doi: 10.1097/ACM.0b013e318217e119. PMID 21512370
- [Result] Cook DA, Hatala R, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hamstra SJ. Technology-enhanced simulation for health professions education: a systematic review and meta-analysis. JAMA. 2011 Sep 7;306(9):978-88. doi: 10.1001/jama.2011.1234. PMID 21900138
- [Result] Norcini JJ, Blank LL, Duffy FD, Fortna GS. The mini-CEX: a method for assessing clinical skills. Ann Intern Med. 2003 Mar 18;138(6):476-81. doi: 10.7326/0003-4819-138-6-200303180-00012. PMID 12639081
- [Result] Norcini JJ, Blank LL, Arnold GK, Kimball HR. The mini-CEX (clinical evaluation exercise): a preliminary investigation. Ann Intern Med. 1995 Nov 15;123(10):795-9. doi: 10.7326/0003-4819-123-10-199511150-00008. PMID 7574198
- [Result] Norcini JJ, Blank LL, Arnold GK, Kimball HR. Examiner differences in the mini-CEX. Adv Health Sci Educ Theory Pract. 1997;2(1):27-33. doi: 10.1023/A:1009734723651. PMID 16180056
- [Result] Hatala R, Ainslie M, Kassen BO, Mackie I, Roberts JM. Assessing the mini-Clinical Evaluation Exercise in comparison to a national specialty examination. Med Educ. 2006 Oct;40(10):950-6. doi: 10.1111/j.1365-2929.2006.02566.x. PMID 16987184
- [Result] Leblanc VR. Review article: simulation in anesthesia: state of the science and looking forward. Can J Anaesth. 2012 Feb;59(2):193-202. doi: 10.1007/s12630-011-9638-8. Epub 2011 Dec 17. PMID 22179792